CLINICAL TRIAL: NCT03234413
Title: Switching Between Different Types of Botulinum Toxin-A in Children With Cerebral Palsy Treated for Spasticity: a Safety Retrospective Evaluation
Brief Title: Safety on Switching Between Different Botulinum Toxin-A
Status: Completed | Type: Observational
Sponsor: Nigar Dursun (Other)
Responsible Party: Sponsor-Investigator, Nigar Dursun, Professor, MD, Kocaeli University
Organization: Kocaeli University (Other)
Other Study IDs: KU GOKAEK 2017/91
Record Dates: First submitted 2017-07-19; First posted 2017-07-31 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy
Keywords: Botulinum Toxin-A
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A
  Other Names: Botox, Dysport

SUMMARY:
Clinical guidelines recommend the use of Botulinum Toxin-A (BoNT-A) for localized/segmental spasticity in children with cerebral palsy. At the Kocaeli University (KOU) Department of Physical Medicine and Rehabilitation (PMR) more than 800 patients have been injected with the two approved toxinA types; OnabotulinumtoxinA or AbobotulinumtoxinA.

With this study investigators would like to evaluate retrospectively if switching from one toxin to another is safe as well as to evaluate if the efficacy when switching from one toxin to another was maintained.

DETAILED DESCRIPTION:
A data base was designed to capture all data that were considered relevant to the treatment evaluation. The data were transcribed directly from participants medical records. For the purpose of the study, data from the two subsequent visits where a different type of toxin was given will be collected and evaluated . In order to collect the pre and post status in terms of safety and efficacy, for each participant, data corresponding to the 6 previous and posterior months after the switch of the toxin will also be collected or data corresponding to the previous and posterior visit after the switch of the toxin will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosis of cerebral palsy with respect to Rosenbaum criteria,
* children having received repeated injections with two different types of toxinA treatment into their lower limb(s)

Exclusion Criteria:

* children without repeated Botulinum toxin type A injections
* children having received repeated injections with same type of toxinA

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: No active study treatment will be given as this will be a retrospective study. Information on children with at least two subsequent injection of two different types of toxinA for the treatment of spasticity will be collected and analysed
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Occurence of treatment related adverse events | Up to 30 months
  Overall and per injection cycle

SECONDARY OUTCOMES:
Modified Ashworth Scale | Up to 30 months
  Spasticity Assessment Scale
Tardieu Scale | Up to 30 months
  Spasticity Assessment Scale
Observational Gait Scale | Up to 30 months
  Gait Assessment Scale

OTHER OUTCOMES:
Goal Attainment Scale | Up to 30 months
  Outcome measure for goal selection and goal scaling

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Dursun, MD, Study Director — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No